CLINICAL TRIAL: NCT03201250
Title: A Phase I/II Study of the c-Met Inhibitor Cabozantinib as a Targeted Strategy to Reverse Resistance to the Proteasome Inhibitor Carfilzomib in Refractory Multiple Myeloma
Brief Title: Cabozantinib as a Targeted Strategy to Reverse Carfilzomib Resistance in Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Phase I response to treatment was not as expected and the myeloma field in treatment has changed since initiating the study, so investigators felt the study should not be pursued into Phase II.
Sponsor: University of Nebraska (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0434-17-FB
Record Dates: First submitted 2017-06-19; First posted 2017-06-28 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Multiple Myeloma; Refractory Multiple Myeloma; Relapsed/Refractory Multiple Myeloma
Keywords: carfilzomib; cabozantinib; proteasome inhibitor; resistance
MeSH Terms: conditions — Multiple Myeloma | interventions — cabozantinib; carfilzomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Combination of cabozantinib, carfilzomib and dexamethasone
  Cabozantinib: patients will receive cabozantinib orally once daily continuously during the four weeks of a 28-day cycle.
  Carfilzomib: carfilzomib will be administered intravenously over 10 minutes, on two consecutive days, each week for three weeks (Days 1, 2, 8, 9, 15, and 16), followed by a 12-day rest period (Days 17 to 28). Each 28-day period is considered one treatment cycle.
  Dexamethasone: dexamethasone will be administered at 40 mg orally or intravenously on days 1, 8,15 and 22 of each 28-day cycle (for patient age ≥ 75, acceptable to be given as 20 mg orally or intravenously on days 1, 2, 8, 9, 15, 16, 22, 23)
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib:
  Phase I: Level -1 = 20 mg or Level 0 = 40 mg or Level +1 = 60 mg, PO daily on days 1-28 Phase II: One of phase I dosing levels identified as MTD, PO daily on days 1-28
  Carfilzomib: 27 mg/m2 IV over 10 min on days 1, 2, 8, 9, 15, 16
  Dexamethasone: 40 mg PO/IV on days 1, 8,15 and 22 (for patient age ≥ 75, acceptable to be given as 20 mg PO/IV on days 1, 2, 8, 9, 15, 16, 22, 23)
  Other Names: carfilzomib; dexamethasone

SUMMARY:
In the currently proposed phase I/II study, the investigators aim to treat patients with relapsed and/or relapsed refractory Multiple Myeloma who have progressed on carfilzomib-based therapy with an FDA approved c-MET inhibitor, cabozantinib.

DETAILED DESCRIPTION:
In the currently proposed phase I/II study, the investigators aim to treat patients with relapsed and/or relapsed refractory multiple myeloma (MM) who have progressed on carfilzomib-based therapy with an FDA approved c-MET inhibitor, cabozantinib. Our hypothesis is that the additional rescue blockade with cabozantinib added to the carfilzomib will (1) be safe and tolerable and (2) will show activity by demonstrating objective response to combination carfilzomib/cabozantinib therapy. In correlative studies, the investigators aim to show that (1) the serum and marrow MUC20 levels which will be judged by genomic and flow cytometric studies will directly correlate with primary plasma cell MUC20/c-Met pathway activation and inversely correlate with protease inhibitor (PI) resistance; and (2) a correlation of the gene and MUC20 expression profiles of patients with clinical outcomes may confirm the biomarker MUC20 as a predictor of disease sensitivity to PI, and allow future personalization of c-Met-targeted therapies, as well as combination approaches based on c-Met inhibitors.

To be eligible for this study, patients must have been previously diagnosed with histologically or cytologically confirmed symptomatic MM, must have measurable disease and have had at least two, but not more than four prior lines of therapy for their disease, with lines of therapy being separated by the presence of documented disease progression. Additionally, patients eligible will be those who have failed carfilzomib either as a single agent as the last form of therapy, or carfilzomib in combination with dexamethasone, or carfilzomib in combination with revlimid and dexamethasone.

In Phase I of this study the investigators will determine the maximum tolerated dose (MTD) among three doses. Dose limiting toxicities (DLTs) will be based solely on adverse events that occur during cycle 1. The initial dose of cabozantinib for all patients treated on this study will be 20 mg P.O. daily, which is designated dose level -1.

Response assessment will be performed at start and after cycle 2 using the serum and/or urine protein electrophoresis with immunofixation and serum free light chains to assess disease burden. Disease response quality will also be assessed after completion of three cycles of therapy, and then every cycle after that. Bone marrow aspiration and biopsy will be performed after the baseline sampling only to confirm the achievement of a complete remission (CR).

All patients will be closely followed for toxicity from the time of informed consent until 30 days after last administration of study medication. Adverse event and serious adverse events will be followed until baseline or less than or equal to grade 1 levels. Every subject who fulfills all aspects of patient eligibility who receives a partial or complete course of chemotherapy will be evaluable for dose limiting toxicity (DLT).

ELIGIBILITY:
Inclusion Criteria:

1. Previously diagnosed symptomatic multiple myeloma (MM), with all 3 of the following IMWG criteria, except as noted:

   * Clonal bone marrow plasma cells ≥ 10%
   * A monoclonal protein in either serum or urine
   * Evidence of end-organ damage that can be attributed to the underlying plasma cell proliferative disorder (to include one of the following)

     * Hypercalcemia (corrected calcium > 2.75 mmol/L or 11.5 mg/dL); OR
     * Renal insufficiency attributable to myeloma (serum creatinine >1.9 mg/dL); OR
     * Anemia; normochromic, normocytic with a hemoglobin value ≥2 g/dL below the lower limit of normal, or a hemoglobin or <10 g/dL; OR
     * Bone lytic lesions, severe osteopenia or pathologic fractures.
   * Patients with a biopsy-proven plasmacytoma and either a serum or urine monoclonal protein will also be considered to have met the diagnostic criteria for multiple myeloma in the absence of clonal marrow plasmacytosis of ≥ 10%.
   * Patient with bone marrow plasma cells of ≥ 60% or serum free light chain ratio of ≥ 100 will also be considered to have met the diagnostic criteria for multiple myeloma.
2. Patients must have measurable disease, with at least one of the following:

   * Serum monoclonal protein level ≥0.5 g/dL for IgG, IgA, or IgM disease
   * M-protein or total serum IgD ≥0.5 g/dL for IgD disease
   * Urinary M-protein excretion of ≥200 mg over a 24-hour period
   * Involved free light chain level ≥10 mg/dL, with an abnormal free light chain ratio
3. Patients must have had at least 1, but not more than 4 prior lines of therapy for their disease, with lines of therapy separated by the presence of documented disease progression [induction + HD chemotherapy and autologous stem cell transplant (SCT) + maintenance therapy constitutes 1 line, provided no progression]
4. Patients must have failed carfilzomib either as a single agent as the last form of therapy, or carfilzomib in combination with dexamethasone, carfilzomib in combination with revlimid and dexamethasone, carfilzomib in combination with pomalidomide and dexamethasone or carfilzomib in combination with cyclophosphamide and dexamethasone. Patients have to have had very good tolerance to carfilzomib in the context of described regimens, with resolved prior toxicity to grade 1 or better, and no toxicities due to carfilzomib that required dose reductions to less than 27 mg/m².
5. Patients must have disease that has relapsed after carfilzomib therapy, with progressive disease being defined as an increase of 25% from the lowest response value in any one or more of the following:

   * Serum M-component (the absolute increase must be ≥0.5 g/dL) and/or
   * Urine M-component (the absolute increase must be ≥200 mg/24 hours) and/or
   * Only in patients without a measurable serum and urine M protein level: the difference between involved and uninvolved FLC levels (absolute increase) must be >10 mg/dL
   * Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
   * Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to the plasma cell proliferative disorder

   Patients with relapsed disease will be considered to be those who have had progression, as defined above, off of any therapy, and who completed their therapy more than 60 days prior to the finding of progression. Patients with relapsed and refractory disease will be considered to be those who have had progression, as defined above, while still on their last line of therapy, or who progressed within 60 days of finishing their most recent therapy.
6. Patients must have completed their most recent drug therapy directed at MM in the following time frames:

   * Chemotherapy, biological therapy, immunotherapy, monoclonal antibody or an investigational therapy at least 3 weeks prior to starting cabozantinib
   * Corticosteroids at least 3 weeks prior to starting cabozantinib, except for a dose equivalent to dexamethasone of ≤4 mg/day
   * Nitrosoureas, nitrogen mustards, mitomycin C at least 6 weeks prior to starting cabozantinib
   * Autologous SCT or chimeric antigen receptor (CAR) T cell therapy at least 12 weeks prior to starting cabozantinib
   * Allogeneic SCT or CAR T cell at least 24 weeks prior to starting cabozantinib, and these patients must also not have moderate to severe active acute or chronic graft versus host disease
7. Patients must be age 19 or older (state of NE)
8. Eastern Cooperative Oncology Group performance status of 0, 1, or 2 Karnofsky ≥60%
9. Patients must have evidence of adequate bone marrow reserves, as defined by the following:

   * ANC ≥1,000 cells/mm3 without growth factors within 1 week of the initiation of treatment
   * Total WBC ≥2,000 cells/mm3 without growth factors within 1 week of the initiation of treatment
   * Hemoglobin ≥8 g/dL without red blood cell transfusions within 2 weeks of the initiation of treatment
   * Platelet counts of ≥100,000 cells/mm3 for patients who have bone marrow plasmacytosis of <50%, or ≥50,000 cells/mm3 for patients who have bone marrow plasmacytosis of ≥50%
10. Patients must have evidence of adequate hepatic function, as defined by the following:

    * Total bilirubin ≤1.5 times the upper limit of the institutional normal values
    * Total AST and ALT ≤2.5 times the upper limit of the institutional normal values
11. Patients must have evidence of adequate renal function, as defined by the following:

    * Serum creatinine within the institutional normal limits, OR if the creatinine is elevated
    * Creatinine clearance (CrCl) ≥30 mL/min., as measured by a 24-hour urine collection, or estimated by the Cockcroft and Gault formula

    Any patient with urinary protein (otherwise unrelated to urinary myeloma associated M-protein) with excretion > 3.5 g/day will be considered to have developed nephrotic-range proteinuria, and will be taken off study.
12. Patients must have evidence of adequate cardiac function, as defined by the following:

    * Absence of NYHA class II, III, or IV congestive heart failure
    * Absence of uncontrolled angina or hypertension defined as sustained blood pressure > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
    * Absence of the following in the previous 6 months:

      * myocardial infarction;
      * unstable angina pectoris;
      * clinically-significant cardiac arrhythmias defined as grade 3 or 4 according to NCI CTCAE, version 4.0
      * stroke (including transient ischemic attack, or other ischemic event);
      * thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter (eg, vena cava filter) are not eligible for this study)
    * Absence of history of congenital long QT syndrome
13. Patients who have received radiation therapy (RT) must have completed this at least 4 weeks prior to starting therapy with cabozantinib, with the following exceptions:

    * Local RT to enhance bone healing of a pathologic fracture within 2 weeks prior to starting cabozantinib
    * Local RT for post-fracture pain that is refractory to analgesics within 2 weeks prior to starting cabozantinib
14. Patients who have undergone any recent major surgery within 4 weeks prior to starting therapy with cabozantinib, with the following exceptions:

    * Vertebroplasty and/or kyphoplasty must have been within 1 week prior to starting cabozantinib
    * Planned elective surgery unrelated to the patient's diagnosis of MM, such as hernia repair, may be allowed, at the discretion of the principle investigator, as long as it was performed within 2 weeks prior to starting cabozantinib, and patients have recovered fully.
15. HIV seropositive patients with acceptable organ function who meet the patient selection criteria, and who are not on combination antiretroviral therapy, and whose absolute CD4+ count is ≥400 cells per mm3 will be eligible (HIV positive patients on combination antiretroviral therapy will be ineligible)
16. Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (eg, male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s)
17. Female subjects of childbearing potential must not be pregnant at screening. Female patients must be either postmenopausal, free from menses for ≥2 years, surgically sterilized, or willing to use two adequate barrier methods of contraception to prevent pregnancy, or must agree to abstain from heterosexual activity throughout the study. Female patients of childbearing potential must have a negative serum (bHCG) or urine pregnancy before the first dose of cabozantinib or carfilzomib.
18. Understand and able to willingly provide voluntary written informed consent, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care.

Exclusion Criteria:

1. Patients who are receiving any concurrent investigational agent with known or suspected activity against MM, or those whose adverse events due to agents administered more than 4 weeks earlier have not recovered to grade 0 or 1.
2. Patients who have known CNS involvement with MM
3. Patients who have previously been treated with another agent targeting the MUC20/c-Met axis, including either monoclonal antibodies to MUC20 or c-Met, or small molecule inhibitors of c-Met.
4. Patients with a known history of allergic reactions attributed to compounds of similar chemical or biologic composition to cabozantinib.
5. Chronic concomitant treatment with strong CYP3A4 inhibitors (eg, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's Wort) should be avoided because it may significantly decrease cabozantinib concentrations. If patients are taking any strong CYP3A4 inhibitors, alternate medications with no or minimal CYP3A4 inhibitors should be sought prior to trial enrollment.
6. Uncontrolled or ongoing/active infection, or patients with the following history: recent history of hemorrhage or hemoptysis; dehiscence or wound healing complications requiring medical intervention; severe hypertension that cannot be controlled (blood pressure of > 150 systolic or > 100 diastolic mm) with anti-hypertensive therapy within 7 days of first dose of therapy.
7. Pregnant or lactating women
8. Patients with non-secretory MM, active plasma cell leukemia, defined as either having 20% of peripheral WBC comprised of CD138+ plasma cells, or an absolute plasma cell count of 2 x 109/L, known amyloidosis, or known POEMS syndrome
9. Patients who have required plasmapheresis and exchange less than 2 weeks prior to initiation of therapy with cabozantinib
10. Patients with known moderate or severe hepatic impairment, active hepatitis A, B, and/or C infection
11. Patients with a "currently active" second malignancy, other than non-melanoma skin cancer and carcinoma in situ of the cervix. Patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for >5 years, and are considered by their physician to be at less than 30% risk of relapse. Also, patients with basal cell carcinoma of the skin, superficial carcinoma of the bladder, carcinoma of the prostate with a current PSA value of <0.5 ng/mL, or cervical intraepithelial neoplasia are eligible. Patients who are on hormonal therapy for a history of either prostate or breast cancer may enroll, if there has been no evidence of disease progression during the previous 3 years.
12. Allergy to carfilzomib or cabozantinib or any excipients
13. Uncontrolled intercurrent illness including medical, psychiatric, cognitive or other conditions, psychiatric illness/social situations that would compromise the patient's ability to understand the patient information, to give informed consent, to comply with the study protocol or to complete the study or, in the judgment of the Principal Investigator, would make the patient inappropriate for study participation.
14. The subject has experienced any of the following:

    * clinically-significant GI bleeding within 6 months before the first dose of study treatment;
    * GI disorders particularly those associated with a high risk of perforation or fistula formation including:

      * Tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
      * Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before randomization,
    * hemoptysis of ≥ 0.5 teaspoon (2.5 ml) of red blood within 3 months before the first dose of study treatment;
    * any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment.
15. The subject has radiographic evidence of cavitating pulmonary lesion(s);
16. The subject has tumor invading or encasing any major blood vessels;
17. The subject has evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib;
18. QTcF > 500 msec within 1 month before the first dose of study treatment:

    - Three ECGs must be performed for eligibility determination. If the average of these three consecutive results for QTcF is ≤ 500 msec, the subject meets eligibility in this regard.
19. Inability to swallow intact tablets
20. The subject has PT/INR or PTT test ≥ 1.3 x the laboratory ULN within 7 days before the first dose of study treatment;
21. Concomitant anticoagulation at therapeutic doses with oral anticoagulants (eg, warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (eg, clopidogrel);
22. Subjects who have Carfilzomib-related posterior reversible encephalopathy syndrome (PRES) and thrombotic microangiopathy (TMA) should not be challenged with Carfilzomib.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhamed Baljevic, MD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated prior to starting the Phase II portion of the study.
Groups:
- Level -1 = 20 mg: Combination of cabozantinib, carfilzomib and dexamethasone
  Cabozantinib: patients will receive cabozantinib orally once daily continuously during the four weeks of a 28-day cycle.
  Cabozantinib:
  Phase I: Level -1 = 20 mg
  Carfilzomib: 27 mg/m2 IV over 10 min on days 1, 2, 8, 9, 15, 16
  Dexamethasone: 40 mg PO/IV on days 1, 8,15 and 22 (for patient age ≥ 75, acceptable to be given as 20 mg PO/IV on days 1, 2, 8, 9, 15, 16, 22, 23)
- Level 0 = 40 mg: Combination of cabozantinib, carfilzomib and dexamethasone
  Cabozantinib: patients will receive cabozantinib orally once daily continuously during the four weeks of a 28-day cycle.
  Cabozantinib:
  Phase I: Level 0 = 40 mg
  Carfilzomib: 27 mg/m2 IV over 10 min on days 1, 2, 8, 9, 15, 16
  Dexamethasone: 40 mg PO/IV on days 1, 8,15 and 22 (for patient age ≥ 75, acceptable to be given as 20 mg PO/IV on days 1, 2, 8, 9, 15, 16, 22, 23)
- Level +1 = 60 mg: Combination of cabozantinib, carfilzomib and dexamethasone
  Cabozantinib: patients will receive cabozantinib orally once daily continuously during the four weeks of a 28-day cycle.
  Cabozantinib:
  Phase I: Level +1 = 60 mg
  Carfilzomib: 27 mg/m2 IV over 10 min on days 1, 2, 8, 9, 15, 16
  Dexamethasone: 40 mg PO/IV on days 1, 8,15 and 22 (for patient age ≥ 75, acceptable to be given as 20 mg PO/IV on days 1, 2, 8, 9, 15, 16, 22, 23)
Period: Overall Study
Arm/Group | Level -1 = 20 mg | Level 0 = 40 mg | Level +1 = 60 mg
Started | 8 | 3 | 0
Completed | 5 | 3 | 0
Not Completed | 3 | 0 | 0
Not completed — screen failures | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We only included the 8 subjects that passed eligibility and were dosed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Level -1 = 20 mg | Level 0 = 40 mg | Level +1 = 60 mg | Total
Number analyzed (Participants) | 5 | 3 | 0 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 1 | 2 |  | 3
  >=65 years | 4 | 1 |  | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 |  | 3
  Male | 3 | 2 |  | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 1 | 0 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 2 |  | 2
  White | 4 | 1 |  | 5
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Daily Cabozantinib Given
Description: The investigators will study three dose levels using the 3+3 algorithm. MTD will be assess with dose limiting toxicities (DLTs) based solely on adverse events that occur during cycle 1.
Time Frame: 1 cycle (approximately 28 days)
Population: Only subjects that were dosed are included in this analysis
Measure: Number; unit: mg
Groups:
- Treatment: Combination of cabozantinib, carfilzomib and dexamethasone Cabozantinib: patients will receive cabozantinib orally once daily continuously during the four weeks of a 28-day cycle.
  Cabozantinib:
  Phase I: Level -1 = 20 mg or Level 0 = 40 mg or Level +1 = 60 mg, PO daily on days 1-28 Carfilzomib: 27 mg/m2 IV over 10 min on days 1, 2, 8, 9, 15, 16 Dexamethasone: 40 mg PO/IV on days 1, 8,15 and 22 (for patient age ≥ 75, acceptable to be given as 20 mg PO/IV on days 1, 2, 8, 9, 15, 16, 22, 23)
Arm/Group | Treatment
Number analyzed (Participants) | 8
mg | 20

2. Primary Outcome: Overall Response Rate (ORR)
Description: Per International Myeloma Working Group (IMWG) Uniform Response Criteria guidelines as assessed by laboratory blood tests: Complete Response (CR), negative immunofixation of serum and urine, disappearance of soft tissue plasmacytomas, <5% plasma cells in bone marrow; Stringent Complete Response (sCR), same as CR plus normal serum free light chain (FLC) ratio and absence of clonal plasma cells; Very Good Partial Response (VGPR), serum and urine M-component still detectable by immunofixation or >/= 90% reduction in serum M-component plus a urine M component of, 100mg per 24hrs; Partial Response (PR) ≥ 50% reduction of the serum M-protein and 24 hour urinary M-protein by ≥ 90%, or to < 200 mg per 24 hours. If serum and urine M-protein are not measurable, a ≥ 50% decrease in the difference between involved and uninvolved FLC levels is required OR If FLC is also not informative, ≥ 50% reduction in bone marrow plasma. ORR includes following only: CR+sCR+VGPR+PR
Time Frame: 2 cycles (approximately 56 days)
Population: Two subjects were not included in this analysis as the protocol states that an individual must complete at least 2 cycles before a best response (ORR) could be established.
Measure: Count of Participants; unit: Participants
Arm/Group | Level -1 = 20 mg | Level 0 = 40 mg | Level +1 = 60 mg
Number analyzed (Participants) | 3 | 3 | 0
Participants | 1 | 0 | 0

3. Secondary Outcome: Response Durability Assessed by Progression Free Survival (PFS)
Description: Progressive Disease (PD) is defined per International Myeloma Working Group (IMWG) Uniform Response Criteria guidelines is an increase of 25% from the lowest response value in any one or more of the following: Serum M-component and/or Urine M-component and/or in patients without a measurable serum and urine M protein level: the difference between involved and uninvolved FLC levels must be >10mg/dL, Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing lesions or plasmacytomas, Development of hypercalcemia attributed solely to the plasma cell proliferative disorder
Time Frame: variable, defined by individual response durability in individual patients who would stay on therapy until disease progression
Population: No subjects were dosed at 60 mg dose level.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Level -1 = 20 mg | Level 0 = 40 mg | Level +1 = 60 mg
Number analyzed (Participants) | 5 | 3 | 0
weeks | 25 [12 to 68] | 19 [12 to 28] |

ADVERSE EVENTS:
Time Frame: All patients will be closely followed for toxicity from the time of informed consent until 30 days after last administration of study medication upto approximately 2 years.
Description: Since no subjects were enrolled into the 60 mg dose level for the study number of participants at risk for SAEs, All-Cause Mortality and Other AEs is zero for the dose level +1 = 60mg Arm/Group.
Groups:
- Dose Level -1 = 20 mg: Combination of cabozantinib, carfilzomib and dexamethasone
  Cabozantinib: patients will receive cabozantinib orally once daily continuously during the four weeks of a 28-day cycle.
  Carfilzomib: carfilzomib will be administered intravenously over 10 minutes, on two consecutive days, each week for three weeks (Days 1, 2, 8, 9, 15, and 16), followed by a 12-day rest period (Days 17 to 28). Each 28-day period is considered one treatment cycle.
  Dexamethasone: dexamethasone will be administered at 40 mg orally or intravenously on days 1, 8,15 and 22 of each 28-day cycle (for patient age ≥ 75, acceptable to be given as 20 mg orally or intravenously on days 1, 2, 8, 9, 15, 16, 22, 23)
  Cabozantinib: Cabozantinib:
  Phase I: Level -1 = 20 mg PO daily on days 1-28
  Carfilzomib: 27 mg/m2 IV over 10 min on days 1, 2, 8, 9, 15, 16
  Dexamethasone: 40 mg PO/IV on days 1, 8,15 and 22 (for patient age ≥ 75, acceptable to be given as 20 mg PO/IV on days 1, 2, 8, 9, 15, 16, 22, 23)
- Dose Level 0 = 40 mg: Combination of cabozantinib, carfilzomib and dexamethasone
  Cabozantinib: patients will receive cabozantinib orally once daily continuously during the four weeks of a 28-day cycle.
  Carfilzomib: carfilzomib will be administered intravenously over 10 minutes, on two consecutive days, each week for three weeks (Days 1, 2, 8, 9, 15, and 16), followed by a 12-day rest period (Days 17 to 28). Each 28-day period is considered one treatment cycle.
  Dexamethasone: dexamethasone will be administered at 40 mg orally or intravenously on days 1, 8,15 and 22 of each 28-day cycle (for patient age ≥ 75, acceptable to be given as 20 mg orally or intravenously on days 1, 2, 8, 9, 15, 16, 22, 23)
  Cabozantinib: Cabozantinib:
  Phase I: Level 0 = 40 mg PO daily on days 1-28
  Carfilzomib: 27 mg/m2 IV over 10 min on days 1, 2, 8, 9, 15, 16
  Dexamethasone: 40 mg PO/IV on days 1, 8,15 and 22 (for patient age ≥ 75, acceptable to be given as 20 mg PO/IV on days 1, 2, 8, 9, 15, 16, 22, 23)
- Dose Level +1= 60 mg: Combination of cabozantinib, carfilzomib and dexamethasone
  Cabozantinib: patients will receive cabozantinib orally once daily continuously during the four weeks of a 28-day cycle.
  Carfilzomib: carfilzomib will be administered intravenously over 10 minutes, on two consecutive days, each week for three weeks (Days 1, 2, 8, 9, 15, and 16), followed by a 12-day rest period (Days 17 to 28). Each 28-day period is considered one treatment cycle.
  Dexamethasone: dexamethasone will be administered at 40 mg orally or intravenously on days 1, 8,15 and 22 of each 28-day cycle (for patient age ≥ 75, acceptable to be given as 20 mg orally or intravenously on days 1, 2, 8, 9, 15, 16, 22, 23)
  Cabozantinib: Cabozantinib:
  Phase I: Level +1 = 60 mg, PO daily on days 1-28
  Carfilzomib: 27 mg/m2 IV over 10 min on days 1, 2, 8, 9, 15, 16
  Dexamethasone: 40 mg PO/IV on days 1, 8,15 and 22 (for patient age ≥ 75, acceptable to be given as 20 mg PO/IV on days 1, 2, 8, 9, 15, 16, 22, 23)
Arm/Group | Dose Level -1 = 20 mg | Dose Level 0 = 40 mg | Dose Level +1= 60 mg
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 2/3 | 0/0
Other Adverse Events (participants affected / at risk) | 3/5 | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level -1 = 20 mg (N=5) | Dose Level 0 = 40 mg (N=3) | Dose Level +1= 60 mg (N=0)
Other - Bacteremia infection (Infections and infestations) | 0 (0) | 1 (1) | NA
hypertension (Vascular disorders) | 0 (0) | 1 (1) | NA
hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | NA
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level -1 = 20 mg (N=5) | Dose Level 0 = 40 mg (N=3) | Dose Level +1= 60 mg (N=0)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
hypertension (Vascular disorders) | 2 (2) | 2 (2) | NA
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | NA
platelet count decreased (Investigations) | 0 (0) | 1 (4) | NA
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | NA
alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | NA
aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT03201250/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT03201250/ICF_001.pdf